CLINICAL TRIAL: NCT03007095
Title: Preterm Birth and Social Cognition: of the Executive Functions and Parental Anxiety's Stakes
Brief Title: Preterm Birth and Social Cognition
Acronym: TERM-COG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PO16068*
Record Dates: First submitted 2016-12-27; First posted 2017-01-02 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2023-10

CONDITIONS: Preterm Children

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preterm children (Experimental)
  Interventions: Behavioral: Evaluation of the children's social cognitive development
- term children (Active Comparator)
  Interventions: Behavioral: Evaluation of the children's social cognitive development

INTERVENTIONS:
Behavioral: Evaluation of the children's social cognitive development — standardized neuropsychological tests

SUMMARY:
The study aims at investigating social cognition outcomes of children born prematurely. Social cognition can be briefly defined as a process which underlines people's social and emotional behaviors. There are behavioral and cognitive evidences indicating that preterm children have executive dysfunctions. Executive functions refer to multiple cognitive processes that contribute to human higher order abilities, such as purposeful and future-orientated behavior. The literature regarding development of term born children indicates that executive functions are linked to the emergence of social cognition. Then, the investigators asked if children born prematurely, as they commonly present executive dysfunctions, would show an atypical development of social cognition. Additionally, as it has been shown that parental anxiety is a key factor of preterm children development, the investigators assumed that it should play a role in social cognition outcomes.

DETAILED DESCRIPTION:
The present study examines the social cognition development of very preterm children at 7 to 10 years old. In the literature, there has yet to be any research on social cognition of children born prematurely while preterm children are usually described as having difficulties in social relations. The main hypothesis is that preterm children would present a deficit or a delay in the social cognition development in comparison with that of matched term children, and that this deficit or delay should be explained by executive dysfunctions and parental anxiety.

Social cognition can be defined as the ability to understand the mind of other people and more specifically to perceive emotion, to have empathy, to attribute false-belief, to understand intended meaning, among others. In this study, the investigators will mainly focus on the ability of 80 very preterm children to understand the mind of others, well known as theory of mind in the literature, thanks to small stories involving the thinking and feelings of characters.

The executive functioning, which refers to multiple processes underlying human higher order abilities, will be assessed thanks to standardized neuropsychological tests. In this study, the investigators will focus on the three main well known executive functions: inhibition, working memory and shifting. They expect, consistently with the literature, that preterm children will have executive dysfunctions, and that these will be linked to children theory of mind abilities.

Finally, given that parental anxiety affects child development, the investigators plan to assess some psychological features of children's parents in our study, such the level of parental anxiety. They assume that this level will also be linked to theory of mind abilities of children.

ELIGIBILITY:
Inclusion Criteria:

Preterm children:

* Girls or boys born before 37 weeks of gestational age.
* Aged between 7 to 10 years-old
* At school

Term children:

* Girls or boys born after 37 weeks of gestational age.
* Aged between 6 and 10 years-old: 6 year-olds were included for the mental age matching with preterm children.
* At school

Exclusion Criteria:

* Children :

  * Child with a intrauterine growth failure
  * Child from multiple births
  * Child with organic malformation
  * Child with a genetic anomaly
  * Child with a neuromoteur pathology
  * Child with a global developmental delay (Intellectual quotient inferior to 80).
* Parents :

  * Minor parent (less than 18 year old)
  * Parent with an intellectual disability
  * Parent with a psychotic syndrome
  * Parent who does not understand French

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Social cognition / Theory of mind | Day 0
  small stories involving the thoughts and feelings of characters
working memory | Day 0
  Executives functions
shifting | Day 0
  Executives functions
Trait Anxiety Inventory | Day 0
  Parent's psychological features
Beck Depression Inventory | Day 0
  Parent's psychological features
Social Support Questionnaire | Day 0
  Parent's psychological features
Trauma | Day 0
  Parent's psychological features
Parental Stress Index | Day 0
  Parent's psychological features

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

REFERENCES:
- [Result] Eutrope J, Novo A, Barbe C, Loron G, Rolland AC, Caillies S. Impact of Executive Functions and Parental Anxiety on the Development of Social Cognition in Premature Children: A Cross-Sectional Case-Control Protocol. Front Psychiatry. 2021 Sep 9;12:484571. doi: 10.3389/fpsyt.2021.484571. eCollection 2021. PMID 34566706